CLINICAL TRIAL: NCT05618405
Title: The Effect of General Anaesthesia and Surgery on Sleep-wake Timing in Children: the CLOCKS Kids Observational Study
Brief Title: Changes in Circadian Rhythm After Anaesthesia in Children
Acronym: CLOCKSkids
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jorinde Polderman, Pediatric Anesthesiologist, principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W22_068
Record Dates: First submitted 2022-04-13; First posted 2022-11-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Circadian Rhythm Sleep Disorder; Circadian Rhythm Disorder Caused by Drug; Circadian Rhythm Sleep Disorder, Jet Lag Type; Jet Lag; Anesthesia; Sleep; Sleep Disorders, Circadian Rhythm; Sleep Disturbance
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Jet Lag Syndrome; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children who undergo anesthesia because of surgery: Children, aged between 1-11 years, who undergo general anesthesia because of surgery.
- Children who undergo anesthesia because of an MRI: Children, aged between 1-11 years, who undergo general anesthesia because of an MRI.

SUMMARY:
In this study the investigators will examine the effect of general anesthesia and surgery on sleep duration and sleep quality in children, using questionnaires and a sleep diary.

DETAILED DESCRIPTION:
Objective:

The primary objective is to assess the effect of general anaesthesia and surgery on sleep duration (chronotype) and sleep quality in children aged 1-11 years in the first week after surgery.

Secondary objectives are to determine the duration of the effect of general anaesthesia on chronotype and sleep quality. Furthermore, the investigators will examine factors which may be of influence on the quality and duration of sleep, like postoperative emergence delirium, admission to the hospital, Face, Legs, Activity, Cry, Consolability scale (FLACC) / Numeric Rating Scale (NRS) scores, preoperative sedative medication and postoperative sedative medication.

Study procedures:

Possible participants will be identified on the anaesthetic pre-operative assessment clinic and asked if they object to a phone call with information about research. If not, a researcher will contact the parents by telephone to inform them about the study. After oral consent by both parents, an invitation to fill in the questionnaires will be sent to the parents together with a consent form. Informed consent by both parents will be obtained. Questionnaires can be completed online or on paper, depending on the parents' preference.

Questionnaires:

* Sleep quality: Child's Sleep Habits Questionnaire (CSHQ) on day 3 preoperative and on day 7 postoperative.
* Chronotype: Children's chronotype questionnaire on day 3 preoperative
* Daily sleep diary starting from 3 days preoperative until 7 days postoperative

The following items will be extracted from the electronic health record:

* Demographic criteria: age, gender, type of procedure
* Admission dates
* Preoperative sedative medication
* Postoperative sedative medication
* NRS/FLACC scores during hospital stay All items will be entered in an electronic database (CASTOR)

Primary endpoint The diurnal phase shift the night after surgery, measured by comparing the midpoint of sleep three nights before surgery (as measured by the sleeping log) with midpoint of sleep the night after surgery.

Secondary endpoints

* Change in sleep quality as measured with the CSHQ questionnaire
* Incidence of postoperative sleep problems as measured with the CSHQ questionnaire
* Difference in sleep problems, sleep duration and sleep quality between children who had anaesthesia for magnetic resonance imaging and children who had anaesthesia and surgery
* Influence of pain and sedative medication on sleep duration and quality

ELIGIBILITY:
Inclusion criteria:

* General anaesthesia for surgery or magnetic resonance imaging (MRI) with a minimal duration of 30 minutes
* Age 1-11 years
* Informed consent of both parents

Exclusion criteria:

* Parents are not fluent in Dutch
* Known severe sleep disturbances
* Postoperative admission to paediatric intensive care unit
* Moderate to severe developmental disorder (IQ<85)
* American Society of Anesthesiologists (ASA) classification > 3

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-11 years planned for elective surgery or a procedure requiring general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The diurnal phase shift | Baseline (1wk before anesthesia) - First night post-anesthesia
  The diurnal phase shift the night after surgery, measured by comparing the midpoint of sleep three nights before surgery (as measured by the sleeping log) with midpoint of sleep the night after surgery.

SECONDARY OUTCOMES:
Change in sleep quality | 3 days pre-anaesthesia - 7 days post-anaesthesia
  The change in subjective sleep quality, including incidence of sleep problems (e.g. sleepwalking, nightmares), as measured by the Children's Sleep Habits Questionnaire (CSHQ), between the month prior to 3 nights pre-anesthesia and 1 week post-anesthesia. This is measured on a likert scale 1 meaning no sleep problems and 5 meaning a lot of sleep problems. The answers from questionnaire 1 (3 days preoperative) are compared to answers of questionnaire 2 (7 days postoperative)
Changes in all sleep times | 3 days pre-anaesthesia - 7 days post-anaesthesia
  Changes in all sleep parameters (i.e. sleep on- and offset times, sleep duration, sleep latency) when comparing baseline (as measured by the Children's ChronoType Questionnaire (CCTQ) 3 days pre-anesthesia) to all 10 nights of the sleeping log.
Difference in sleep quality between children who had anaesthesia for magnetic resonance imaging and children who had anaesthesia and surgery | 3 days pre-anaesthesia - 7 days post-anaesthesia
  Difference in subjective sleep quality (as measured by the CSHQ) between patients receiving anesthesia for magnetic resonance imaging and patients receiving anesthesia for a surgical procedure. Answers are on a likerts scale with 1 meaning no sleep problems and 5 meaning a lot of sleep problems.
Difference in sleep-wake timing | 3 days pre-anaesthesia - 7 days post-anaesthesia
  Difference in changes in sleep-wake timing (as measured by the sleeping log, units are minutes) between patients receiving anesthesia for magnetic resonance imaging and patients receiving anesthesia for a surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hermanides, Prof, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, locatie AMC, Amsterdam, North Holland, Netherlands